CLINICAL TRIAL: NCT05224960
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled Trial to Evaluate the Efficacy and Safety of Human Umbilical Cord-derived Mesenchymal Stem Cells in the Treatment of Decompensated Cirrhosis Patients(MSC-DLC-2)
Brief Title: Human Umbilical Cord-derived Mesenchymal Stem Cells for Decompensated Cirrhosis (MSC-DLC-2)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing 302 Hospital (Other)
Collaborators: Chinese PLA General Hospital (Other); Shanghai Changzheng Hospital (Other); LanZhou University (Other); Jin Yin-tan Hospital (Unknown); Hainan Hospital of Chinese PLA General Hospital (Unknown); Vcanbio Cell and Gene Engineering Corp., Ltd. (Industry); Third Affiliated Hospital, Sun Yat-Sen University (Other); Xinjiang Kashi Area Number 1 Hospital (Unknown)
Responsible Party: Principal Investigator, Fu-Sheng Wang, Head of Treatment and Research Center for Infectious Diseases, Principle Investigator, Clinical Professor, Beijing 302 Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MSC-DLC-2
Record Dates: First submitted 2022-01-26; First posted 2022-02-04 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Decompensated Cirrhosis

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, multicenter study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Human Umbilical Cord-Mesenchymal Stem Cells (UC-MSCs) (Experimental): UC-MSCs plus standard of care (SOC).
  Interventions: Biological: UC-MSCs
- Placebo (Placebo Comparator): Placebo plus SOC.
  Interventions: Biological: Placebo(solution without UC-MSCs)

INTERVENTIONS:
Biological: UC-MSCs — 3 doses of UC-MSCs intravenously at day 1, day 8, day 15.
  Arms: Human Umbilical Cord-Mesenchymal Stem Cells (UC-MSCs)
Biological: Placebo(solution without UC-MSCs) — 3 doses of placebo intravenously at day 1, day 8, day 15.
  Arms: Placebo

SUMMARY:
Decompensated cirrhosis has a high overall mortality rate. There is a large unmet need for safe and alternative therapeutic potions. This clinical trial is to inspect the efficiency and safety of mesenchymal stem cells (MSCs) therapy for decompensated cirrhosis.

DETAILED DESCRIPTION:
Decompensated cirrhosis has a high overall mortality rate. Liver transplantation is still the most effective treatment for decompensated cirrhosis. However, the shortage of matched liver sources, high costs, and rejection after liver transplantation restrict the development of liver transplantation.

Mesenchymal stem cells (MSC) are a kind of pluripotent stem cells belonging to mesoderm, which mainly exist in connective tissue and organ interstitium. At present, MSC can be isolated and prepared from bone marrow, fat, synovium, bone, muscle, lung, liver, pancreas and amniotic fluid and umbilical cord blood . Due to its wide range of sources and self-proliferation and differentiation ability, MSCs have therapeutic potential for many diseases, including acute and chronic liver diseases.

In recent years, our team has carried out a series of clinical trials using umbilical cord-derived MSCs to treat patients with end-stage liver disease, decompensated cirrhosis, primary biliary cholangitis, and status after liver transplantation and found that MSCs therapy can significantly improve patient liver function, reduce post-transplantation rejection, reduce complications, improve quality of life, and improve survival. Other investigators have also found in clinical trials with MSCs from different sources that treatment with MSCs can improve MELD scores or liver function levels to varying degrees. However, some studies have found no significant difference between the treatment group and the control group, and MSCs may differentiate into hepatic stellate cells and have the risk of promoting liver fibrosis, it is believed that MSCs do not favor the improvement of liver function in these studies. Therefore, the therapeutic effects of MSCs need to be further validated by larger multicenter randomized controlled clinical trials.

The investigators will do a prospective, double-blind, muliticenter, randomised trial to assess treatment with three intravenous doses of MSCs compared with placebo. 140 decompensated cirrhosis patients will be recruited in China. 70 patients will receive i.v. transfusion 3 times of MSCs and the standard of care as the treated group. In addition, the 70 patients will receive placebo and standard of care as control group.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to provide written informed consent;
2. Aged 18 to 75 years (including 18 and 75 years), male or female;
3. Patients diagnosed with decompensated liver cirrhosis based on clinical findings, laboratory tests, imaging findings and/or representative pathological findings (decompensated liver cirrhosis is defined as the occurrence of at least one serious complication, including esophageal and gastric varices bleeding, hepatic encephalopathy, ascites, spontaneous bacterial peritonitis and other serious complications);
4. The Model for End-stage Liver Disease (MELD) score 15 to 30 points.

Exclusion Criteria:

1. Appearance of active variceal bleeding, overt hepatic encephalopathy (HE), refractory ascites or hepatorenal syndrome within 1 month prior to screening visit.
2. Uncontrolled severe infection within 2 weeks of screening.
3. Patients with hepatitis B virus-related decompensated liver cirrhosis may discontinue antiviral therapy during the study, or those who with antiviral therapy for HBV for less than 12 months, or hepatitis B virus (HBV) DNA ≥ detection limit at the time of screening.
4. Patients with hepatitis C virus-related decompensated liver cirrhosis may discontinue antiviral therapy during the study, or those who with antiviral therapy for HCV for less than 12 months, or hepatitis C virus (HCV) RNA ≥ detection limit at the time of screening (except HCV RNA< detection limit without any antiviral treatment).
5. Patients under treatment with corticosteroids for autoimmune hepatitis for less than 6 months.
6. Trans-jugular intrahepatic portosystemic shunts (TIPS) insertion within 6 months prior to study inclusion.
7. Active drinkers with alcohol-related decompensated cirrhosis are unwilling to stop alcohol abuse after inclusion.
8. Significant renal insufficiency (serum creatinine ≥ 1.2 times upper normal limit); Severe electrolyte abnormality (serum sodium level < 125 mmol/L); Severe leukopenia (white blood cell count < 1 × 10E9/L).
9. Patients with biliary obstruction, or portal vein spongiosis.
10. Patients with surgical history such as splenic cut-off flow.
11. Patients with malignant tumors within 5 years, except those with basal cell carcinoma, squamous cell carcinoma and/or carcinoma in situ who had received curative treatment and curative resection.
12. Patients with a prior history of major organ transplantation or complicated with significant disease of heart, lung, kidney, blood, endocrine and other systems.
13. Drug abuse, drug dependence and patients who receive methadone treatment or with psychosis.
14. Against the human immunodeficiency virus antibody (Anti - HIV) or syphilis antibody test results were positive.
15. Pregnancy, lactation or with recent fertility plan during the test and 6 months after the test.
16. Highly allergic, or have a history of severe allergies, known severe allergies to the investigational drug or any of the excipients.
17. History of pulmonary embolism.
18. Patients who had previously received stem cell therapy or were intolerant to cell therapy.
19. The proposed line of liver transplants within three months.
20. Participants in other clinical trials within the last 3 months.
21. Any other clinical condition which the investigator considers would make the patient unsuitable for the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2025-06-27 (Estimated); Study Completion 2027-06-20 (Estimated)

PRIMARY OUTCOMES:
Change in Model for End-Stage Liver Disease (MELD) score from baseline to 28th day | Baseline, 28th day
  The Model for End-stage Liver Disease (MELD) is a scoring system that evaluates the liver function reserve and prognosis of patients with chronic liver disease by creatinine, international normalized ratio (INR), and bilirubin-conjugated cirrhosis etiology.

SECONDARY OUTCOMES:
Change in MELD score from baseline to 24 months | up to 24 months
Incidence of each complication associated with decompensated cirrhosis | up to 24 months
Liver transplant-free survival | month 12 and 24
Incidence of liver failure | month 12 and 24
plasma albumin (ALB) | up to 24 months
plasma prealbumin (PALB) | up to 24 months
total bilirubin (TBIL) | up to 24 months
serum cholinesterase (CHE) | up to 24 months
prothrombin activity (PA) | up to 24 months
Child-Turcotte-Pugh (CTP) score | up to 24 months
  Child-Turcotte-Pugh (CTP) score is a scoring system that evaluates the liver function.
EuroQol Group 5-Dimension Self-Report Questionnaire (EQ-5D) | up to 24 months
ChronicLiver Disease Questionnaire (CLDQ) | up to 24 months
Incidence of liver cancer | up to 24 months
Incidence of Treatment-Emergent Adverse Events and Serious Adverse Events | up to 24 months
Alanine Aminotransferase (ALT) | up to 24 months
Aspartate Aminotransferase (AST) | up to 24 months
Alkaline Phosphatase (ALP) | up to 24 months
Gamma-Glutamyl transferase (GGT) | up to 24 months
plasma ammonia | up to 24 months
international normalized ratio (INR) | up to 24 months
creatinine （Cr） | up to 24 months
Prothrombin time (PT) | up to 24 months
Liver transplant-free survival rate | month 12 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Sheng Wang, MD, PhD, Study Chair — Beijing 302 Hospital
Locations (7):
- China (7):
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Third Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Hainan hospital of Chinese PLA General Hospital, Sanya, Hainan
  - Jin Yin-tan Hospital, Wuhan, Hubei
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - Xinjiang Kashi Area Number 1 Hospital, Kashgar, Xinjiang
  - Beijing 302 Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Yes
After approval from the steering committee and the Human Genetic Resources Administration of China, this trial data can be shared with qualifying researchers who submit a proposal with a valuable research question. A contract should be signed.